CLINICAL TRIAL: NCT00887341
Title: Phase II Multi-centre, Randomized, Parallel Group, Pilot Trial to Compare the Incidence of Tocilizumab Related Infusion Reactions in Moderate to Severe RA Patients When Infusion is Made Over 1 Hour Against 31 Minutes
Brief Title: A Study Comparing Infusion Rates of Tocilizumab in Patients With Moderate to Severe Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML22254; 2008-006443-39
Record Dates: First submitted 2009-04-22; First posted 2009-04-23 (Estimated); Results first posted 2014-10-22 (Estimated); Last update posted 2014-10-22 (Estimated); Status verified 2014-10

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]
- 2 (Active Comparator)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv every 4 weeks for 6 infusions; first infusion 1h duration, subsequent infusions 31 minutes duration
  Arms: 1
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv every 4 weeks for 6 infusions; each infusion 1h duration
  Arms: 2

SUMMARY:
This 2 arm study will compare the incidence of tocilizumab-related infusion reactions, using 2 different infusion times, in patients with moderate to severe rheumatoid arthritis who have shown an inadequate response to DMARDs (Disease Modifying Anti Rheumatic Drugs) or anti-TNFs.Patients will be randomized to one of 2 groups, to receive tocilizumab 8mg/kg iv every 4 weeks either a)over a 1h infusion time for all administrations or b) a 1h infusion time for the first administration, followed by a 31 minute infusion time for subsequent administrations (unless drug-related infusion reactions occur).The anticipated time on study treatment is 3-12 months, and the target sample size is <100 individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult patients, >=18 years of age;
* active moderate or severe rheumatoid arthritis;
* active disease for >6 months;
* inadequate response to a stable dose of non-biologic DMARDs or antiTNFs.

Exclusion Criteria:

* rheumatic autoimmune disease other than rheumatoid arthritis;
* prior history of, or current inflammatory joint disease other than rheumatoid arthritis;
* major surgery (including joint surgery) within 8 weeks prior to screening, or planned major surgery within 6 months following enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2009-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (21):
- Spain (21):
  - Vitoria-Gasteiz, Alava
  - Villajoyosa, Alicante
  - Ávila, Avila
  - Menorca, Balearic Islands
  - Palma de Mallorca, Balearic Islands
  - Badalona, Barcelona
  - L'Hospitalet de Llobregat, Barcelona
  - Mollet del Vallès, Barcelona
  - Torrelavega, Cantabria
  - Castellon, Castellon
  - Alcalá de Henares, Madrid
  - Madrid, Madrid
  - San Sebastián de los Reyes, Madrid
  - Vigo, Pontevedra
  - Gijón, Principality of Asturias
  - Oviedo, Principality of Asturias
  - Alzira, Valencia
  - San Juan, Valencia
  - Valenica, Valencia
  - Galdakao, Vizcaya
  - Zaragoza, Zaragoza

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab, 1 Hour Infusions: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) via intravenous (IV) infusion (over 1 hour), once every 4 weeks for 6 infusions (up to 24 weeks).
- Tocilizumab, 31 Minute Infusions: Participants received tocilizumab 8 mg/kg via IV infusion, once every 4 weeks for 6 infusions (up to 24 weeks). The first infusion was 1 hour; the remaining 5 infusions were administered over a period of 31 minutes as long as no infusion reactions occurred. If an infusion reaction occurred, 1 hour infusions were used for all subsequent remaining infusions.
Period: Overall Study
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Started | 37 | 39
Completed | 35 | 36
Not Completed | 2 | 3
Not completed — Refused treatment | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) Population: all participants enrolled in the study who had been randomly assigned to one of the two study treatments and received at least one dose of study drug.
Groups:
- Tocilizumab, 1 Hour Infusions: Participants received tocilizumab 8 mg/kg via IV infusion (over 1 hour), once every 4 weeks for 6 infusions (up to 24 weeks).
- Total: Total of all reporting groups
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions | Total
Number analyzed (Participants) | 37 | 39 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.65 (12.71) | 52.46 (10.47) | 52.55 (11.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 28 | 63
  Male | 2 | 11 | 13

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With an Infusion Reaction Within 24 Hours After Infusion
Description: An infusion reaction was defined as any adverse event (AE) that occurred during the infusion or during the 24 hours following the infusion.
Time Frame: Screening, Baseline, and Weeks 4, 8, 12, 16, 20, and 24
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants | 29.7 | 17.9
Statistical Analysis 1: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Test type: Superiority or Other; p = 0.238, Chi-squared

2. Secondary Outcome: Percentage of Participants Discontinuing Tocilizumab in Response to an AE or Serious AE (SAE)
Time Frame: Weeks 4, 8, 12, 16, 20 and Final Visit
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants | 2.7 | 0.0

3. Secondary Outcome: Percentage of Participants Discontinuing Tocilizumab for Any Reason
Time Frame: Weeks 4, 8, 12, 16, 20 and Final Visit
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants | 2.7 | 2.6

4. Secondary Outcome: Percentage of Participants With a Reduction of at Least 1.2 Units on the Disease Activity Scale Based on 28-Joint Count (DAS28) by Visit
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28-joint count, the erythrocyte sedimentation rate (ESR) (millimeters per hour [mm/hr]) and Patient's Global Assessment of Disease (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 less than or equal to (≤)3.2 equals (=) low disease activity, DAS28 greater than (>)3.2 to 5.1 = moderate to high disease activity; DAS28 less than (<) 2.6 = remission. A reduction of at least 1.2 units was considered a clinically significant difference.
Time Frame: Weeks 4, 8, 12, 16, 20 and Final Visit
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants
  Week 4 | 56.7 | 61.9
  Week 8 | 58.6 | 74.1
  Week 12 | 77.8 | 92.3
  Week 16 | 88.5 | 88.0
  Week 20 | 88.9 | 84.0
  Final visit | 80.8 | 91.7

5. Secondary Outcome: Percentage of Participants Achieving a DAS28 Score <3.2 by Visit
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hr), and Patient's Global Assessment of Disease (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 ≤3.2=low disease activity, DAS28 >3.2 to 5.1=moderate to high disease activity; DAS28 <2.6=remission.
Time Frame: Weeks 4, 8, 12, 16, 20 and Final Visit
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants
  Week 4 | 22.2 | 32.0
  Week 8 | 25.0 | 60.0
  Week 12 | 46.9 | 77.1
  Week 16 | 59.4 | 77.1
  Week 20 | 68.8 | 79.4
  Final visit | 64.3 | 80.6

6. Secondary Outcome: Percentage of Participants Achieving a DAS28 Score <2.6 (Remission)
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hr) and Patient's Global Assessment of Disease (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 ≤3.2=low disease activity, DAS28 >3.2 to 5.1=moderate to high disease activity; DAS28 <2.6=remission.
Time Frame: Weeks 4, 8, 12, 16, 20 and Final Visit
Population: ITT population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants
  Week 4 | 11.1 | 20.0
  Week 8 | 18.8 | 34.3
  Week 12 | 34.4 | 57.1
  Week 16 | 40.6 | 51.4
  Week 20 | 56.3 | 58.8
  Final visit | 46.4 | 74.2

7. Secondary Outcome: DAS28 Score by Visit
Description: DAS28 calculated from the number of swollen joints and tender joints using the 28-joint count, the ESR (mm/hr) and Patient's Global Assessment of Disease (participant-rated arthritis activity assessment) with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity. DAS28 ≤3.2=low disease activity, DAS28 >3.2 to 5.1=moderate to high disease activity; DAS28 <2.6=remission. Last observation carried forward (LOCF) visit took the last non-missing post-baseline available value.
Time Frame: Weeks 4, 8, 12, 16, 20, and Final Visit
Population: ITT Population; n (number)=number of participants analyzed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 38
units on a scale
  Baseline visit (n=36,38) | 5.75 (1.18) | 5.32 (1.14)
  Week 4 (n=36,25) | 4.28 (1.33) | 3.62 (1.27)
  Week 8 (n=32,35) | 4.14 (1.54) | 3.05 (1.20)
  Week 12 (n=32,35) | 3.30 (1.32) | 2.66 (1.04)
  Week 16 (n=32,35) | 3.07 (1.50) | 2.64 (1.18)
  Week 20 (n=32,34) | 2.78 (1.33) | 2.41 (1.22)
  Final visit (n=28,31) | 2.72 (1.40) | 2.19 (1.06)
  LOCF visit (n=37,38) | 2.92 (1.56) | 2.37 (1.13)

8. Secondary Outcome: Percentage of Participants Achieving American College of Rheumatology 20 Percent (%) Improvement (ACR20 Response)
Description: ACR20 response defined as an improvement of ≥20% in swollen joint count (SJC; 66 joints) and tender joint count (TJC; 68 joints) as well as ≥20% improvement in at least 3 of the following 5 remaining ACR assessments: Patient Global Assessment of Pain; Patient Global Assessment of Disease Activity; Physician Global Assessment of Disease Activity; Health Assessment Questionnaire - Disability Index (HAQ-DI); and acute phase reactive factors (ESR or C-Reactive Protein [CRP])
Time Frame: Weeks 4, 8, 12, 16, 20 and Final Visit
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants
  Week 4 | 26.5 | 48.5
  Week 8 | 51.5 | 59.4
  Week 12 | 60.0 | 69.7
  Week 16 | 74.2 | 60.6
  Week 20 | 81.8 | 54.5
  Final visit | 70.6 | 64.7
Statistical Analysis 1: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 4; Test type: Superiority or Other; p = 0.121, Chi-squared
Statistical Analysis 2: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 8; Test type: Superiority or Other; p = 0.809, Chi-squared
Statistical Analysis 3: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 12; Test type: Superiority or Other; p = 0.367, Chi-squared
Statistical Analysis 4: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 16; Test type: Superiority or Other; p = 0.339, Chi-squared
Statistical Analysis 5: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 20; Test type: Superiority or Other; p = 0.017, Chi-squared
Statistical Analysis 6: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Final visit; Test type: Superiority or Other; p = 0.451, Chi-squared

9. Secondary Outcome: Percentage of Participants Achieving ACR 50% Improvement (ACR50 Response)
Description: ACR50 response defined as an improvement of ≥50% in SJC (66 joints) and TJC (68 joints) as well as ≥50% improvement in at least 3 of the following 5 remaining ACR assessments: Patient Global Assessment of Pain; Patient Global Assessment of Disease Activity; Physician Global Assessment of Disease Activity; HAQ-DI; and acute phase reactive factors (ESR or CRP).
Time Frame: Weeks 4, 8, 12, 16, 20 and Final Visit
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants
  Week 4 | 11.4 | 20.6
  Week 8 | 26.5 | 39.4
  Week 12 | 35.5 | 47.1
  Week 16 | 53.1 | 45.5
  Week 20 | 65.6 | 45.5
  Final visit | 54.5 | 45.7
Statistical Analysis 1: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 4; Test type: Superiority or Other; p = 0.377, Chi-squared
Statistical Analysis 2: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 8; Test type: Superiority or Other; p = 0.387, Chi-squared
Statistical Analysis 3: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 12; Test type: Superiority or Other; p = 0.304, Chi-squared
Statistical Analysis 4: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 16; Test type: Superiority or Other; p = 0.509, Chi-squared
Statistical Analysis 5: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 20; Test type: Superiority or Other; p = 0.110, Chi-squared
Statistical Analysis 6: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Final visit; Test type: Superiority or Other; p = 0.504, Chi-squared

10. Secondary Outcome: Percentage of Participants Achieving ACR 70% Improvement (ACR70 Response)
Description: ACR70 response defined as an improvement of ≥70% in SJC (66 joints) and TJC (68 joints) as well as ≥70% improvement in at least 3 of the following 5 remaining ACR assessments: Patient Global Assessment of Pain; Patient Global Assessment of Disease Activity; Physician Global Assessment of Disease Activity; HAQ-DI; and acute phase reactive factors (ESR or CRP).
Time Frame: Weeks 4, 8, 12, 16, 20 and Final Visit
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants
  Week 4 | 0.0 | 2.9
  Week 8 | 12.1 | 14.7
  Week 12 | 22.6 | 28.6
  Week 16 | 25.1 | 28.6
  Week 20 | 33.3 | 29.4
  Final visit | 38.2 | 30.6
Statistical Analysis 1: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 4; Test type: Superiority or Other; p = 0.327, Chi-squared
Statistical Analysis 2: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 8; Test type: Superiority or Other; p = 0.786, Chi-squared
Statistical Analysis 3: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 12; Test type: Superiority or Other; p = 0.482, Chi-squared
Statistical Analysis 4: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 16; Test type: Superiority or Other; p = 0.680, Chi-squared
Statistical Analysis 5: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 20; Test type: Superiority or Other; p = 0.690, Chi-squared
Statistical Analysis 6: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Final Visit; Test type: Superiority or Other; p = 0.516, Chi-squared

11. Secondary Outcome: Percentage of Participants Achieving ACR 90% Improvement (ACR90 Response)
Description: ACR90 response defined as an improvement of ≥90% in SJC (66 joints) and TJC (68 joints) as well as ≥90% improvement in at least 3 of the following 5 remaining ACR assessments: Patient Global Assessment of Pain; Patient Global Assessment of Disease Activity; Physician Global Assessment of Disease Activity; HAQ-DI; and acute phase reactive factors (ESR or CRP).
Time Frame: Weeks 4, 8, 12, 16, 20 and Final Visit
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants
  Week 4 | 0.0 | 0.0
  Week 8 | 2.9 | 2.9
  Week 12 | 3.1 | 5.7
  Week 16 | 3.0 | 11.1
  Week 20 | 8.8 | 5.7
  Final visit | 12.1 | 11.1
Statistical Analysis 1: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 8; Test type: Superiority or Other; p = 0.970, Chi-squared
Statistical Analysis 2: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 12; Test type: Superiority or Other; p = 0.587, Chi-squared
Statistical Analysis 3: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 16; Test type: Superiority or Other; p = 0.184, Chi-squared
Statistical Analysis 4: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Week 20; Test type: Superiority or Other; p = 0.600, Chi-squared
Statistical Analysis 5: Comparison: Tocilizumab, 1 Hour Infusions vs Tocilizumab, 31 Minute Infusions; Final Visit; Test type: Superiority or Other; p = 0.937, Chi-squared

12. Secondary Outcome: C-Reactive Protein (CRP) Levels
Description: CRP is an inflammation marker. High levels of this protein indicate inflammation in diseases such as Rheumatoid Arthritis. CRP is measured in milligrams per liter (mg/L).
Time Frame: Screening, Baseline, Weeks 4, 8, 12, 16, 20, and Final Visit
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 38
mg/L
  Screening (n=35,38) | 9.28 (9.64) | 10.76 (11.88)
  Baseline (n=30,35) | 11.49 (15.39) | 13.68 (26.21)
  Week 4 (n=37,37) | 6.45 (13.52) | 4.29 (8.16)
  Week 8 (n=34,37) | 4.84 (10.98) | 1.93 (2.84)
  Week 12 (n=33,36) | 2.94 (5.80) | 1.78 (3.95)
  Week 16 (n=35,38) | 2.81 (6.86) | 2.08 (4.00)
  Week 20 (n=34,36) | 1.97 (2.52) | 2.66 (7.89)
  Final visit (n=31,34) | 5.42 (13.27) | 2.26 (4.57)

13. Secondary Outcome: Erythrocyte Sedimentation Rate
Description: ESR is an acute phase reactant measured in mm/hr. Reduction in ESR indicates improvement.
Time Frame: Baseline, Weeks 2, 4, 8, 12,16, 20, and 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 37
mm/hr
  Screening (n=37,37) | 37.70 (25.19) | 31.19 (18.62)
  Baseline (n=30,30) | 42.53 (28.60) | 30.40 (17.78)
  Week 4 (n=36,29) | 15.03 (16.16) | 11.41 (8.93)
  Week 8 (n=33,36) | 15.36 (17.06) | 8.67 (8.82)
  Week 12 (n=32,35) | 12.19 (16.63) | 6.77 (6.47)
  Week 16 (n=33,36) | 11.97 (15.39) | 6.50 (6.22)
  Week 20 (n=33,34) | 13.83 (19.91) | 6.29 (6.76)
  Final visit (n=30,33) | 12.00 (13.77) | 6.70 (5.59)

14. Secondary Outcome: HAQ-DI Score by Visit
Description: HAQ-DI is a self-reported, valid assessment of functional disability in rheumatoid arthritis. Assessment based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. HAQ-DI scores range: 0-3: without any difficulty=0, with some difficulty=1, with much difficulty=2, unable to do=3. HAQ-DI total scores expressed as overall mean score with range 0-3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; more than 1=significant functional limitation.
Time Frame: Baseline, Weeks 2, 4, 8, 12, 16, 20 and 24
Population: ITT Population; n=number of participants assessed for the specified parameter at a given visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 38
units on a scale
  Baseline (n=37,37) | 1.6 (0.7) | 1.4 (0.7)
  Week 4 (n=37,37) | 1.4 (0.7) | 1.0 (0.6)
  Week 8 (n=35,37) | 1.3 (0.8) | 0.9 (0.7)
  Week 12 (n=31,36) | 1.1 (0.7) | 0.8 (0.6)
  Week 16 (n=33,38) | 1.0 (0.8) | 0.8 (0.6)
  Week 20 (n=35,37) | 1.0 (0.7) | 0.8 (0.7)
  Final visit (n=35,35) | 0.9 (0.8) | 0.8 (0.7)

15. Secondary Outcome: Percentage of Participants With Improvement of at Least 0.22 in HAQ-DI
Description: HAQ-DI is a self-reported, valid assessment of functional disability in rheumatoid arthritis. Assessment based on ability of participants to perform daily activities in 8 categories: dressing, arising, eating, walking, reaching, gripping, hygiene, and carrying out daily activities. HAQ-DI scores range: 0-3: without any difficulty=0, with some difficulty=1, with much difficulty=2, unable to do=3. HAQ-DI total scores expressed as overall mean score with range 0-3: 0-0.25=normal functioning; 0.25-0.5=mild functional limitation; 0.5-1=moderate functional limitation; more than 1=significant functional limitation. An improvement of 0.22 units in HAQ-DI was considered to be a clinically significant improvement.
Time Frame: Weeks 4, 8, 12, 16, 20 and Final Visit
Population: ITT Population
Measure: Number; unit: percentage of participants
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Number analyzed (Participants) | 37 | 39
percentage of participants
  Week 4 | 48.6 | 48.6
  Week 8 | 62.9 | 54.3
  Week 12 | 64.5 | 58.8
  Week 16 | 72.7 | 52.8
  Week 20 | 68.6 | 54.3
  Final visit | 68.6 | 61.8

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of Screening until the End of Study (24 Weeks)
Arm/Group | Tocilizumab, 1 Hour Infusions | Tocilizumab, 31 Minute Infusions
Serious Adverse Events (participants affected / at risk) | 2/37 | 2/39
Other Adverse Events (participants affected / at risk) | 30/37 | 26/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab, 1 Hour Infusions (N=37) | Tocilizumab, 31 Minute Infusions (N=39)
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Crohn's Disease (Gastrointestinal disorders) | 1 | 0
Hepatitis (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab, 1 Hour Infusions (N=37) | Tocilizumab, 31 Minute Infusions (N=39)
Anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukopenia (Blood and lymphatic system disorders) | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2
Conjunctival hyperaemia (Eye disorders) | 1 | 0
Eye pruritus (Eye disorders) | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Anal fistula (Gastrointestinal disorders) | 1 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 1
Odynophagia (Gastrointestinal disorders) | 1 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 1
Discomfort (General disorders) | 0 | 1
Face oedema (General disorders) | 1 | 0
Temperature intolerance (General disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 1
Bronchitis (Infections and infestations) | 1 | 1
Cellulitis (Infections and infestations) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 2 | 5
Oral herpes (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 2
Respiratory tract infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 2 | 2
Viral infection (Infections and infestations) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 1
Aspiration joint (Investigations) | 0 | 1
Blood cholesterol increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 0
Transaminase increased (Investigations) | 2 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Haemarthrosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Amnesia (Nervous system disorders) | 1 | 0
Aphonia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 4 | 0
Headache (Nervous system disorders) | 1 | 2
Sciatica (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Depressed mood (Psychiatric disorders) | 1 | 0
Depression (Psychiatric disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 0 | 1
Menstrual disorder (Reproductive system and breast disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sneezing (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Dyshidrosis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 1 | 0
Dental implantation (Surgical and medical procedures) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.